CLINICAL TRIAL: NCT04547101
Title: A Single-arm, Open-label, Multicenter, Phase II Study of AK104, a PD-1/CTLA-4 Bispecific Antibody, in Subjects With Locally Advanced Unresectable or Metastatic Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) Solid Tumors
Brief Title: A Study of AK104 in Subjects With Locally Advanced Unresectable or Metastatic MSI-H/dMMR Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to difficuty of erollment and consideration of clinical guideline,The sponsor decided to stop study.
Sponsor: Akeso (Industry)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-205
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: MSI-H/dMMR Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 (Experimental)
  Interventions: Drug: AK104

INTERVENTIONS:
Drug: AK104 — AK104，6 mg/kg IV，every 2 weeks (Q2W)

SUMMARY:
It is a single-arm, open-label, multicenter, phase II study to evaluate the safety, efficacy, pharmacokinetics (PK) and immunogenicity of AK104 as a single agent in subjects with previously-treated locally advanced unresectable or metastatic MSI-H or dMMR solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Have signed written informed consent form voluntarily.
* Male or female, age ≥ 18 years on the day of signing informed consent form.
* ECOG of 0 or 1.
* Estimated life expectancy of ≥3 months.
* Histologically or cytologically documented locally advanced unresectable or metastatic solid tumors.
* Confirmed MSI-H/dMMR status by the central laboratory.
* Have experienced documented disease progression during or after at least first-line therapy.
* Have radiologically measurable disease based on RECIST 1.1.
* Adequate organ function.
* Have agreed to take effective contraception from the date of signing the informed consent form until 120 days after the last administration.

Exclusion Criteria:

* Prior use of investigational products or devices within 4 weeks prior to C1D1 (Cycle 1 Day 1, the first dose of study drug).
* Presence of active autoimmune disease that have received systematic treatment in the past 2 years; or that is judged to be possibly relapsed or requires planned treatment by investigators.
* Active inflammatory bowel disease or that required treatment (e.g. Crohn's disease, ulcerative colitis or chronic diarrhea).
* Prior use of systematic corticosteroid (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to C1D1.
* Prior exposure to tumor immunotherapy, such as checkpoint inhibitors (eg. anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody), checkpoint agonists or cellular therapy.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Known presence or history of interstitial lung disease.
* History of gastrointestinal perforation and/or fistula within 6 months prior to C1D1.
* Serious infections within 4 weeks prior to C1D1.
* Known presence of active tuberculosis.
* Known untreated chronic hepatitis B or chronic hepatitis B virus DNA exceeding 1000 IU/ mL or active hepatitis C virus.
* Receipt of recent radiotherapy or anti-tumor treatment within 4 weeks prior to C1D1.
* Presence of meningeal metastasis, spinal cord compression, leptomeningeal disease or central nervous system metastasis, with some exceptions.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria. Hair loss is excluded
* Known history of sever hypersensitivity reaction to other monoclonal antibodies.
* Known history of allergy or hypersensitivity to AK104 or any of its components.
* Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or PR, based on RECIST v1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with confirmed CR, PR, or SD, based on RECIST v1.1
Duration of response (DoR) | Up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from the start of treatment with AK104 until death due to any cause.
Adverse events (AEs) | From first dose of AK104 through to 90 days after last dose of AK104
  Incidences of treatment-emergent adverse events (TEAEs) , treatment-related adverse events (TRAEs) as assessed by CTCAE v5.0
Observed pharmacokinetics (PK) exposure of AK104 | From first dose of AK104 through to 90 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through to 90 days after last dose of AK104
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable ADAs.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No